CLINICAL TRIAL: NCT01824602
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) in Acute Manic Episodes Associated With Bipolar I Disorder in a Double-blind, Fixed Multiple Dose, Randomised, Placebo-controlled,Multicentre Clinical Trial.
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) in Acute Manic Episodes Associated With Bipolar I Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a slow recruitment rate
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-204
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2013-08

CONDITIONS: BIPOLAR I DISORDER
Keywords: BIPOLAR I DISORDER, Eslicarbazepine acetate
MeSH Terms: interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Eslicarbazepine acetate 1800 mg
  Interventions: Drug: Eslicarbazepine acetate 1800 mg
- Group 2 (Experimental): Eslicarbazepine acetate 1200 mg
  Interventions: Drug: Eslicarbazepine acetate 1200 mg
- Group 3 (Experimental): Eslicarbazepine acetate 600 mg
  Interventions: Drug: Eslicarbazepine acetate 600 mg
- Group 4 (Placebo Comparator): Placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine acetate 1800 mg — Eslicarbazepine acetate to be taken orally, was available as 600 mg tablets.
  Other Names: Esl
  Arms: Group 1
Drug: Eslicarbazepine acetate 1200 mg — Eslicarbazepine acetate to be taken orally, was available as 600 mg tablets.
  Other Names: Esl
  Arms: Group 2
Drug: Eslicarbazepine acetate 600 mg — Eslicarbazepine acetate to be taken orally, was available as 600 mg tablets.
  Other Names: Esl
  Arms: Group 3
Drug: Placebo — Placebo sugar pills
  Other Names: Placebo sugar pills
  Arms: Group 4

SUMMARY:
The primary study objective was to evaluate the dose-dependent efficacy of eslicarbazepine acetate administered at doses of 600, 1200, and 1800 mg over a 3-week period, compared with placebo, as therapy in patients with acute mania. The secondary objectives of this study were to a) evaluate the safety and tolerability of eslicarbazepine acetate (BIA 2-093) administered at doses of 600, 1200, and 1800 mg compared with placebo, b) assess the duration to onset of action in the different dose groups, and c) monitor the appearance of depressive symptoms.

DETAILED DESCRIPTION:
This was a phase II, double-blind, fixed multiple dose, randomised, placebo-controlled, multicentre clinical trial in patients with a diagnosis of bipolar I disorder who experienced an acute manic (including mixed) episode. Patients who met the selection criteria at randomisation visit (V) (V2, Day 1) were randomised to 1 of 4 treatment groups: 600, 1200, or 1800 mg eslicarbazepine acetate, or placebo. Patients started the assigned treatment on Day 1 and were followed for up to 3 weeks. On Day 10, patients who showed no improvement were switched to open-label escape therapy with an established antimanic therapy. Patients could have been hospitalized at screening or at any time during the study at the investigator's discretion. Following randomisation (V2, Day 1), patients were assessed on Days 3, 7, 10, 14, 21, 28, and 56, after which they could either enter a recurrence prevention study, or the study drug could be tapered off and they could undergo follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more.
* A documented diagnosis of bipolar I disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria (i.e., 296.0, 296.4 or 296.6).
* Currently displaying an acute manic (including mixed) episode according to the DSM-IV criteria.
* A Young Mania Rating Scale (YMRS) total score of 20 or greater.
* Symptoms of the current manic episode starting within 2 weeks prior to Randomization (V2, Day 1).
* Able to undergo a standard evaluation, including clinical interview, ratings and laboratory studies.
* Signed informed consent form (ICF).
* Post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation. In case of woman of childbearing potential, patient presents a serum pregnancy test consistent with a non-gravid state and will use double-barrier contraception until at least the post-study visit (PSV).

Exclusion Criteria:

* History of schizophrenia or schizoaffective disorder, psychotic features or rapid cycling.
* Currently treated with carbamazepine or oxcarbazepine.
* History of unresponsiveness, intolerance or hypersensitivity to related compounds (carbamazepine, oxcarbazepine or licarbazepine).
* Use of any depot-neuroleptics for the current manic episode
* Abuse of stimulating drugs or use of any systemic sympathicomimetic drug within the previous 2 weeks.
* Electroconvulsive therapy (ECT) within the previous 3 months
* History of dependence or chronic abuse from alcohol, drugs or medications within the last year.
* Judged clinically to be at risk of harm to self or others.
* Second or third-degree atrioventricular blockade not corrected with a pacemaker.
* Relevant ECG or laboratory abnormalities.
* Calculated creatinine clearance <30 ml/min [men: (140-age) x weight / serum creatinine x 72; women: (0.85) (140-age) x weight / serum creatinine x 72. Age in years, weight in kg, and serum creatinine in mg/dl].
* Pregnancy or nursing.
* Participation in other drug clinical trial within the last 2 months before Randomization visit
* Not ensured capability to perform the trial or to comply with the study protocol (e.g. mental retardation or severe inability to communicate);
* Any other uncontrolled clinically relevant disorder.
* Previous treatment with Eslicarbazepine Acetate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrício Soares-da-Silva, MD, PhD, Study Director — BIAL - Portela & Ca. SA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: STUDY DATES: From: 28 Feb 2006 To: 13 Nov 2006 Study centers: 25 study centers in Europe, South Africa and South America: 7 centers in Croatia, 6 centers in Spain, 6 centers in Argentina, 1 center in Chile and 5 centers in South Africa.
Pre-assignment Details: Patients who met the selection criteria at randomisation visit (V) (V2, Day 1) were randomised to 1 of 4 treatment groups: 600, 1200, or 1800 mg eslicarbazepine acetate, or placebo. Patients started the assigned treatment on Day 1 and were followed for up to 3 weeks.
Groups:
- Group 4: Placebo: Placebo pills
  Placebo : Placebo sugar pills
- Group 3: Eslicarbazepine Acetate 600 mg: Eslicarbazepine acetate 600 mg
  Eslicarbazepine acetate 600 mg : Eslicarbazepine acetate to be taken orally, was available as 600 mg tablets.
- Group 2: Eslicarbazepine Acetate 1200 mg: Eslicarbazepine acetate 1200 mg
  Eslicarbazepine acetate 1200 mg : Eslicarbazepine acetate to be taken orally, was available as 600 mg tablets.
- Group 1: Eslicarbazepine Acetate 1800 mg: Eslicarbazepine acetate 1800 mg
  Eslicarbazepine acetate 1800 mg : Eslicarbazepine acetate to be taken orally, was available as 600 mg tablets.
Period: Overall Study
Arm/Group | Group 4: Placebo | Group 3: Eslicarbazepine Acetate 600 mg | Group 2: Eslicarbazepine Acetate 1200 mg | Group 1: Eslicarbazepine Acetate 1800 mg
Started | 11 | 8 | 9 | 10
Safety Population | 11 | 8 | 9 | 10
Intent-to-treat Population | 11 | 8 | 9 | 9
Completed | 10 | 8 | 5 | 5
Not Completed | 1 | 0 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Patient non-compliance | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 2
Not completed — Treatment failure | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 4: Placebo | Group 3: Eslicarbazepine Acetate 600 mg | Group 2: Eslicarbazepine Acetate 1200 mg | Group 1: Eslicarbazepine Acetate 1800 mg | Total
Number analyzed (Participants) | 11 | 8 | 9 | 10 | 38
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 9 | 9 | 37
  >=65 years | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9 | 4 | 22
  Male | 3 | 7 | 0 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Young Mania Rating Scale (YMRS) Total Score From Baseline Until the End of the 3-week Treatment Period
Description: The YMRS is used to assess disease severity in patients who have been previously diagnosed with mania and it has proven psychometric properties through 11 item multiple-choice diagnostic questionnaire and the total score is determined from the summation of each 11 individual scores (and can range from 0 - 60) based on the patient's subjective feedback of his clinical condition over the previous 48 hours. A higher score indicates a worse rating for symptoms related to mania. At every visit throughout the study, investigators administered the YMRS. The results of the primary analysis of efficacy were calculated using Analysis of covariance (ANCOVA) with Last Observation Carried Forward (LOCF). Primary variable is presented through ANCOVA results for absolute change in YMRS total score from baseline (V2) to end of treatment (V7). A responder has at least 50% improvement (reduction) in the YMRS total score or has a total score of less than 12 points at the end of treatment period.
Time Frame: baseline and 3-week
Population: The ITT efficacy population of 37 patients consisted of all randomised patients who received at least one dose of investigational product and at least 1 post-baseline YMRS assessment. If a patient discontinues before the end of the 3-week treatment period then the last observation will be carried forward (LOCF).
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo; ESL 600 mg; ESL 1200 mg: ITT Population
- ESL 1800 mg: (ITT Population
Arm/Group | Placebo | ESL 600 mg | ESL 1200 mg | ESL 1800 mg
Number analyzed (Participants) | 11 | 8 | 9 | 9
units on a scale | -17.7 (7.34) | -16.9 (2.75) | -16.7 (9.11) | -11.3 (10.89)

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Placebo; ESL 600 mg; ESL 1200 mg; ESL 1800 mg: Safety Population
Arm/Group | Placebo | ESL 600 mg | ESL 1200 mg | ESL 1800 mg
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/8 | 0/9 | 1/10
Other Adverse Events (participants affected / at risk) | 7/11 | 4/8 | 9/9 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | ESL 600 mg (N=8) | ESL 1200 mg (N=9) | ESL 1800 mg (N=10)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | ESL 600 mg (N=8) | ESL 1200 mg (N=9) | ESL 1800 mg (N=10)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 5 (5) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other